CLINICAL TRIAL: NCT07053735
Title: An Exploratory Clinical Study of Nimotuzumab in Bladder - Sparing Chemoradiotherapy for Muscle - Invasive Bladder Cancer
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Shangbin QIN, Doctor, Peking University First Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-209
Record Dates: First submitted 2025-06-27; First posted 2025-07-08 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-06

CONDITIONS: Bladder (Urothelial, Transitional Cell) Cancer
Keywords: bladder cancer; TMT; radiation oncology
MeSH Terms: conditions — Neoplasms; Urinary Bladder Neoplasms | interventions — nimotuzumab; Radiotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nim (Experimental)
  Interventions: Drug: Nimotuzumab and Radiotherapy

INTERVENTIONS:
Drug: Nimotuzumab and Radiotherapy — 1. nimotuzumab: 200mg, iv, qw, used for 5 weeks.
  2. radiotherapy: radiotherapy is performed according to clinical routine;

SUMMARY:
The goal of this exploratory study is to evaluate the safety and efficacy of nimotuzumab combined with chemoradiotherapy in bladder - preserving treatment for MIBC patients who are ineligible for or decline radical cystectomy. The main questions it aims to answer are:

Does nimotuzumab combined with radiotherapy reduce adverse events in elderly bladder cancer patients? Does this combination improve objective response rate (ORR), progression - free survival (PFS), overall survival (OS), and bladder preservation rate in these patients? Participants will be MIBC patients treated with nimotuzumab and chemoradiotherapy, with a planned 5 - year follow - up to assess treatment efficacy and safety.

ELIGIBILITY:
Inclusion Criteria:

Signed informed consent. Aged ≥18. Histologically confirmed urothelial carcinoma of the bladder, staged T2a-T4a, anyN, M0, or recurrent T1 high - grade tumors (7th - edition AJCC staging).

Unsuitable or intolerant to cystectomy, or with comorbidities making systemic chemotherapy intolerable, or chemotherapy - averse, or recurrent after prior TURBT and unsuitable for further TURBT or cystectomy.

ECOG performance status 0-2. No severe hematopoietic or major organ dysfunction, or immunodeficiency. Pre - enrollment lab values: white blood cell count ≥3.5×10⁹/L, absolute neutrophil count ≥1.5×10⁹/L, platelets ≥50×10⁹/L, hemoglobin ≥90 g/L; renal: serum creatinine ≤1.2 mg/dL or creatinine clearance ≥60 mL/min; hepatic: total bilirubin ≤3.0×ULN, AST/ALT ≤2.0×ULN; coagulation: INR ≤2.0.

Agreed contraception during the trial for fertile individuals; females of childbearing potential must have a negative pregnancy test within 7 days before initial dosing.

No prior chemotherapy, targeted, or immunotherapy for cancer.

Exclusion Criteria:

Metastatic cancer. Previous pelvic/abdominal radiotherapy. Uncontrolled infection, intractable epilepsy, high intracranial pressure, hypertension, hyperglycemia, angina (Grade 1/symptomatic/≥Grade 2), peripheral neuropathy, or a history of myocardial infarction/heart failure within 6 months, or jaundice due to hepatic insufficiency.

HIV, active hepatitis B (HBsAg and HBV - DNA positive), or active hepatitis C (HCV - RNA positive).

Major surgery within 4 weeks before enrollment. Participation in another clinical trial within 4 weeks before enrollment. Other uncontrolled malignancies within the past 5 years (except cervical in - situ carcinoma, squamous cell skin cancer, or localized basal cell carcinoma).

Any other researcher - identified reason making participation unsuitable.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-06-30 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
ORR | 1 year
PFS | 5 years
OS | 5 years